CLINICAL TRIAL: NCT02841917
Title: Oxidative Stress Response in Patients With Severe Aortic Stenosis Undergoing Transcatheter or Surgical Aortic Valve Replacement (ROS Study)
Brief Title: Reactive Oxygen Species Following Aortic Valve Replacement
Acronym: ROS
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CAR0508
Record Dates: First submitted 2016-07-13; First posted 2016-07-22 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken for measurement of reactive oxygen species
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transcatheter Aortic Valve Replacement: ROS Post TAVR
- Surgical Aortic Valve Replacement: ROS Post SAVR

SUMMARY:
Surgical aortic valve replacement (SVAR) is currently the 'Gold Standard' therapy for patients with severe symptomatic aortic stenosis (AS). Approximately 30-50% of patients with severe AS are deemed inoperable due to comorbidities such as severe respiratory disease, chronic renal disease and peripheral vascular disease. Transcatheter aortic valve replacement (TAVR) has emerged as a novel therapeutic modality for inoperable patients and an effective alternative to SAVR in selected high and intermediate-risk patients. Myocardial ischemia and reperfusion injury (MRI), mediated by reactive oxygen species (ROS), related to cardiopulmonary bypass has been linked to adverse clinical outcomes following cardiac surgery. In contrast to SAVR, transcatheter deployment of aortic prostheses requires shorter time of ischemia and hypotension and may be associated with less ROS mediated MRI. Inflammatory responses and reperfusion injury following TAVR have not been previously described nor compared to SAVR. The aim of this study is therefore to compare the oxidative stress response in patients with isolated severe symptomatic AS undergoing SAVR or TAVR and determine whether it correlates with clinical outcomes.

DETAILED DESCRIPTION:
Myocardial ischemia and reperfusion injury (MRI) related to cardio-pulmonary bypass has been linked to adverse clinical outcomes following cardiac surgery. Changes in ROS following SAVR have been well documented in the literature. Furthermore, pre-operative ROS markers such as malondialdehyde have been shown to be predictors of adverse outcomes after 30-day and 1-year follow-up. In contrast to SAVR, TAVR is associated with shorter duration of myocardial ischemia and hypotension ad may thus be associated with a lower degree of MRI. Inflammatory responses and reperfusion injury following TAVR have not been described nor have they been compared with SAVR.

Cellular respiration leads to the generation of partially reduced oxygen derivatives called ROS. Under normal physiological conditions, ROS serve as integral components of cellular signaling pathways. A balanced redox state is established between the major ROS producing systems (NADPH oxidase, xanthine oxidase, nitric oxide synthase, myeloperoxidase and lipoxygenases) and the major antioxidant systems (catalase, α-tocopherol, ascorbic acid, superoxide dismutase, glutathione peroxidase and glutathione S transferases that conjugate reduced GSH to hydrophobic organic compounds and glutathione). Excess production or reduced degradation of ROS by the antioxidant defense systems imposes an oxidative burden upon the cellular environment leading to modification of numerous biomolecules and functional defects.

In MRI the enzyme xanthine oxidase catalyzes the formation of uric acid with the coproduction of superoxide. Superoxide release results in the recruitment and activation of neutrophils and their adherence to endothelial cells, which stimulates the formation of xanthine oxidase in the endothelium, with further superoxide production. Oxidation of DNA and proteins may then follow leading to membrane damage because of lipid peroxidation leading to alterations in membrane permeability, modification of protein structure and functional changes. Oxidative damage to the mitochondrial membrane can also occur resulting in membrane depolarization and the uncoupling of oxidative phosphorylation with altered cellular respiration. This can ultimately lead to mitochondrial damage, release of cytochrome c, activation of caspases and apoptosis.

Although TAVR may not expose the myocardium to the same level of MRI than SAVR, patients undergoing TAVR have greater numbers of co-morbidities and may thus have a greater baseline ROS burden than patients undergoing SAVR. As the generation of ROS in patients undergoing TAVR and whether differences in ROS levels in such patients correlates with clinical outcomes has not been described. The prospective study will attempt to address both of these questions.

ELIGIBILITY:
Inclusion Criteria:

1. Severe symptomatic aortic stenosis defined as aortic valve area <1 cm2, mean aortic gradient >40 mm Hg or Vmax > 4 m/s amenable for transcatheter or surgical aortic valve replacement.

Exclusion Criteria:

1. Severe comorbidities , advance age, frailty or thoracic anatomy unfavorable for surgical aortic valve replacement.
2. Anatomy precluding transcatheter aortic valve replacement.
3. Requirement for concomitant coronary artery bypass grafting.
4. Requirement for concomitant mitral, tricuspid, or pulmonary valve surgery.
5. Allergy to aspirin or clopidogrel.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic aortic stenosis undergoing transcatheter or surgical aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Ascertain the concentrations of serum isoprostanes, nitrites and sulphides following transcatheter and surgical aortic valve replacement. | 24 hours
  Serum measurements will be undertaken using standard immunoassay techniques.

SECONDARY OUTCOMES:
Ascertain potential differences in the generation of reactive oxygen species that have been outlined in the primary outcomes with cardiovascular mortality. | 30 days clinical follow-up
  Clinical follow-up will be undertaken either by a clinic visit or by telephone contact.
Ascertain potential differences in the generation of reactive oxygen species that have been outlined in the primary outcomes with myocardial infarction. | 30 days clinical follow-up.
  Clinical follow-up will be undertaken either by a clinic visit or by telephone contact.
Ascertain potential differences in the generation of reactive oxygen species that have been outlined in the primary outcomes with stroke. | 30 days clinical follow-up.
  Clinical follow-up will be undertaken either by a clinic visit or by telephone contact.
Ascertain potential differences in the generation of reactive oxygen species that have been outlined in the primary outcomes with major bleeding. | 30 days clinical follow-up.
  Clinical follow-up will be undertaken either by a clinic visit or by telephone contact.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mahmoudi, MD,PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Gabriel Maluenda, MD, Study Director — Centro Cardiovascular, Hospital San Borja, Chile
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Creager MA, Curtis LH, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Stevenson WG, Yancy CW; American College of Cardiology; American College of Cardiology/American Heart Association; American Heart Association. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Thorac Cardiovasc Surg. 2014 Jul;148(1):e1-e132. doi: 10.1016/j.jtcvs.2014.05.014. Epub 2014 May 9. No abstract available. PMID 24939033
- [Result] Bach DS, Siao D, Girard SE, Duvernoy C, McCallister BD Jr, Gualano SK. Evaluation of patients with severe symptomatic aortic stenosis who do not undergo aortic valve replacement: the potential role of subjectively overestimated operative risk. Circ Cardiovasc Qual Outcomes. 2009 Nov;2(6):533-9. doi: 10.1161/CIRCOUTCOMES.109.848259. Epub 2009 Oct 27. PMID 20031890
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Result] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Result] Larmann J, Theilmeier G. Inflammatory response to cardiac surgery: cardiopulmonary bypass versus non-cardiopulmonary bypass surgery. Best Pract Res Clin Anaesthesiol. 2004 Sep;18(3):425-38. doi: 10.1016/j.bpa.2003.12.004. PMID 15212337
- [Result] Scolletta S, Carlucci F, Biagioli B, Marchetti L, Maccherini M, Carlucci G, Rosi F, Salvi M, Tabucchi A. NT-proBNP changes, oxidative stress, and energy status of hypertrophic myocardium following ischemia/reperfusion injury. Biomed Pharmacother. 2007 Feb-Apr;61(2-3):160-6. doi: 10.1016/j.biopha.2006.10.007. Epub 2007 Feb 20. PMID 17350221
- [Result] Cavalca V, Tremoli E, Porro B, Veglia F, Myasoedova V, Squellerio I, Manzone D, Zanobini M, Trezzi M, Di Minno MN, Werba JP, Tedesco C, Alamanni F, Parolari A. Oxidative stress and nitric oxide pathway in adult patients who are candidates for cardiac surgery: patterns and differences. Interact Cardiovasc Thorac Surg. 2013 Dec;17(6):923-30. doi: 10.1093/icvts/ivt386. Epub 2013 Sep 7. PMID 24014619
- [Result] Hausenloy DJ, Yellon DM. The evolving story of "conditioning" to protect against acute myocardial ischaemia-reperfusion injury. Heart. 2007 Jun;93(6):649-51. doi: 10.1136/hrt.2007.118828. PMID 17502643
- [Result] Rodrigo R, Korantzopoulos P, Cereceda M, Asenjo R, Zamorano J, Villalabeitia E, Baeza C, Aguayo R, Castillo R, Carrasco R, Gormaz JG. A randomized controlled trial to prevent post-operative atrial fibrillation by antioxidant reinforcement. J Am Coll Cardiol. 2013 Oct 15;62(16):1457-65. doi: 10.1016/j.jacc.2013.07.014. Epub 2013 Jul 31. PMID 23916928
- [Result] Granger DN. Role of xanthine oxidase and granulocytes in ischemia-reperfusion injury. Am J Physiol. 1988 Dec;255(6 Pt 2):H1269-75. doi: 10.1152/ajpheart.1988.255.6.H1269. PMID 3059826
- [Result] Zimmerman JJ. Defining the role of oxyradicals in the pathogenesis of sepsis. Crit Care Med. 1995 Apr;23(4):616-7. doi: 10.1097/00003246-199504000-00003. No abstract available. PMID 7712748
- [Result] Macdonald J, Galley HF, Webster NR. Oxidative stress and gene expression in sepsis. Br J Anaesth. 2003 Feb;90(2):221-32. doi: 10.1093/bja/aeg034. PMID 12538380